CLINICAL TRIAL: NCT04263376
Title: Can Bariatric Surgery-Induced Shift in Gut Microbiome Protect Against Non-Alcoholic Fatty Liver Disease? A Step Toward Replicating Metabolic Surgery Results Without Surgery
Brief Title: Bariatric Surgery-Induced Shift in Gut Microbiome and NAFLD
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ali Aminian, Associate Professor, The Cleveland Clinic
Other Study IDs: CCF IRB 19-438
Record Dates: First submitted 2019-12-27; First posted 2020-02-10 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; NAFLD
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed as a prospective pilot study for longitudinal assessment of fecal microbiome related to medical and surgical weight loss. The investigators follow the standard of care for perioperative and intraoperative management of study participants. The only addition to the standard of care protocol will be collection of fecal samples at 3 time points. This will enable investigators to compare changes in and effects by microbiota after low-calorie diet versus after bariatric surgery .

ELIGIBILITY:
Inclusion Criteria:

* Be an eligible candidate for bariatric surgery based on standard criteria in place, have been enrolled in bariatric surgery program at Cleveland Clinic Main Campus, and have been cleared and approved for bariatric surgery by the BMI bariatric program and his/her health insurance
* Have a Body Mass Index (BMI) more than 35 kg/m2
* Have type 2 diabetes (T2D) (but not type 1 diabetes, see exclusion criteria) as defined by

  1. If untreated (as per ADA standards of care) FPG > or = 126 mg/dL (7.0 mmol/L). Fasting is defined as no caloric intake for at least 8 h OR 2-h PG > or = 200 mg/dL (11.1 mmol/L) during OGTT. The test should be performed as described by the WHO, using a glucose load containing the equivalent of 75-g anhydrous glucose dissolved in water OR A1C > or = 6.5% (48 mmol/mol). The test should be performed in a laboratory using a method that is NGSP certified and standardized to the DCCT assay OR In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose > or = 200 mg/dL (11.1 mmol/L).
  2. the use of any antidiabetic drug or glucose lowering agent, including biguanides (metformin), thiazolidinediones, alpha-glucosidase inhibitors, sulfonylurea, meglitinides, DPP4-inhibitors, GLP1-agonists, SGLT2i, any type of insulin.
* Have the ability and willingness to participate in the study and agree to the study terms
* As a standard of care, have a negative urine pregnancy test prior to surgery for women of childbearing potential. A woman of childbearing potential is one who is biologically capable of becoming pregnant. This includes women who are using contraceptives or whose sexual partners are either sterile or using contraceptives.

Exclusion Criteria:

* Any contra-indication for bariatric surgery (standard of care)
* Lack of insurance coverage for bariatric surgery
* Diabetes mellitus other than T2D including Type 1 diabetes or Latent Autoimmune Diabetes of the Adult (LADA) as defined by personal history of diabetic ketoacidosis or by positive auto-antibodies to glutamic Acid Decarboxylase (GAD-65), Islet Cell Antibodies (ICA), Insulin Autoantibodies (IAA), or to protein tyrosine phosphatase (IA-2A) Monogenetic or neonatal diabetes
* Prior bariatric surgery of any kind.
* Known history of chronic liver disease except for NAFLD/NASH: hepatitis, positive serologic test result for hepatitis B surface antigen and/or hepatitis C antibody, alpha-1-antitrypsin deficiency.
* Known Gastrointestinal disorders including a known history of celiac disease and/or any other malabsorptive disorders or inflammatory bowel disease (Crohn's disease or ulcerative colitis).
* Psychiatric disorders including dementia, active psychosis, severe depression requiring > 2 medications, history of suicide attempts, alcohol or drug abuse within the previous 12 months.
* Smoking within the previous 3 months.
* Pregnancy.
* Malignancy within five years (except squamous cell and basal cell cancer of the skin). Subjects diagnosed with early / stage 1 cancer that have been successfully treated are eligible per Investigator discretion.
* Use of any medications (prescription or OTC), including herbal or other supplements for treatment of obesity, or liver conditions at the time of consent.
* Any condition or major illness that, in the investigator's judgment, places the subject at undue risk by participating in the study.
* Unable to understand the risks, realistic benefits and compliance requirements of each program.
* Use of investigational therapy or participation in any other clinical trial within 12 weeks prior to signing the ICF.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are in the evaluation process for Roux-en-Y Gastric Bypass (RYGB) and Sleeve Gastrectomy (SG) will be offered the opportunity to volunteer for this study.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in human gut microbiota | 3 months after surgery
  Test for intrapersonal longitudinal changes in human gut microbiota in patients with obesity undergoing bariatric surgery at 3 time points: baseline (preoperative), after diet-induced non-surgical weight loss, and 3-months post-operative.
  Metagenomic characterization of gut microbial communities will be longitudinally examined with human feces at 3 time points. Microbiota profiles will be assessed in fecal samples using V4 variable regions of the 16S rRNA gene by MiSeq 250-base paired-end multiplex sequencing. Moreover, total microbial cell counts in fecal samples will be determined using flow cytometry in order to have a quantitative microbiome profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Aminian, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No